CLINICAL TRIAL: NCT06896370
Title: Risk of Gastric Cancer in High-risk Asymptomatic Carriers of Helicobacter Pylori: an Observational Cohort Study
Brief Title: An Observational Study for Gastric Cancer in Asymptomatic Carriers of High Risk Helicobacter Pylori
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Dazhi Xu, Fudan University
Other Study IDs: 2025observational study
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Gastric (Stomach) Cancer; Helicobacter Infection
MeSH Terms: conditions — Stomach Neoplasms; Helicobacter Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- exposure group: Hp positive + high risk SNP
  Interventions: Other: observational study
- Control 1: Hp positive + non-high risk SNP
  Interventions: Other: observational study
- Control 2: Hp negative
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — By prospectively following a population of asymptomatic carriers carrying high-risk Hp SNP subtypes and non-high-risk subtypes, the incidence of gastric cancer and progression of gastric precancerous lesions were compared between the groups.

SUMMARY:
This study is intended to be a prospective observational cohort study. The incidence of gastric cancer and progression of gastric precancerous lesions will be compared between groups through prospective follow-up of a population of asymptomatic carriers harboring high-risk Hp SNP subtypes and non-high-risk subtypes.

DETAILED DESCRIPTION:
Primary study objective: to assess the difference in the incidence of gastric cancer between asymptomatic carriers of high-risk SNP subtypes of H. pylori and the non-high-risk population during the follow-up period.

Secondary research objectives: 1. To observe and compare the cumulative incidence and progression of gastric precancerous lesions (e.g., atrophic gastritis, intestinal metaplasia, etc.) in each population group during the follow-up period.2. To explore the interaction of high-risk SNPs on the risk of gastric cancer in the context of different age, gender or other risk factors (e.g. diet, smoking, alcohol abuse, family history, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. No previous history of gastric cancer (no radical surgery or radiotherapy treatment for gastric cancer);
3. Able and willing to provide informed consent and willing to accept baseline and follow-up examinations;
4. Able to cooperate in completing HP testing (breath test, gastroscopic biopsy or other standard testing methods) and HP SNP typing by stool testing;
5. No obvious gastric symptoms at the time of initial screening, no progressive gastric cancer or serious gastric diseases (e.g., perforated acute ulcers, upper gastrointestinal hemorrhage, etc.) detected, and no need for urgent surgery (not planned within 3 months) or other therapeutic interventions for the time being.

Exclusion Criteria:

1. Diagnosed gastric cancer or other malignant tumors of the digestive tract;
2. Comorbid serious underlying diseases (e.g., severe cardiopulmonary insufficiency, liver and renal failure, etc.) that are expected to have a short survival time or are not suitable for long-term follow-up;
3. Inability to complete or refusal to undergo HP testing, SNP gene testing or follow-up;
4. Presence of severe mental illness or incapacity for civil behavior that prevents completion of the study;
5. Pregnant or breastfeeding women who are temporarily excluded;
6. Other conditions that the investigator considers unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited mainly from communities in Tongling, Anhui Province.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2035-05-01 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in incidence of gastric cancer (pathologically or imaging-confirmed gastric cancer) between high-risk and non-high-risk groups. | From enrollment to the end of the study in 10 years